CLINICAL TRIAL: NCT04496024
Title: Determination of a Trough Serum Concentration of Ofloxacin Associated to Increase in Side Effects Frequency in Elderly Treated for Bone and Joint Infection
Brief Title: Ofloxacin Concentration-toxicity Relationship in the Elderly
Acronym: ROSCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2019_843_0018
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Ofloxacin; Bone and Joint Infection; Therapeutic Drug Monitoring; Adverse Drug Reactions
Keywords: ofloxacin; Bone and Joint Infection; therapeutic drug monitoring; Adverse Drug Reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Ofloxacin; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: ofloxacin — ofloxacin treatment in patients with bone and joint infections
Other: questionnaire — questionnaire of ofloxacine side effects will be completed by the clinician at Day 3, Day 21 and Day 42
Biological: Ofloxacin Serum concentration — Serum concentration of ofloxacin will be measured at Day 3 (Cmin and Cmax), Day 21 and Day 42 (Cmin).

SUMMARY:
Ofloxacin is a gold standard antibiotic for the treatment of bone and joint infections due to sensible staphylococcus strains. However, in the elderly, inter-individual variability of the pharmacokinetics may reduce the efficacy or increase toxicity. The occurrence of ofloxacin side effects is likely to be increased in case of higher exposition. However, the serum concentration-toxicity relationship has not yet been determined. The purpose of this project is to assess the association between the residual serum concentration of ofloxacin at day 3 and the occurrence of at least one adverse effect attributable to ofloxacin, and determine a threshold toxicity concentration if this association exists.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 65 years hospitalized at the University Hospital of Amiens for an uncomplicated bone and joint infections
* Indication for oral switch to ofloxacin

Exclusion Criteria:

* Patient refusing to participate in the study
* Patient under guardianship or curators or deprived of public rights
* Any liver or biliary injury
* Any contraindications to ofloxacin

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of one adverse reaction attributable to ofloxacin in patients with bone and joint infections | day 3
  Frequency of at least one adverse reaction attributable to ofloxacin in patients with bone and joint infections

CONTACTS AND LOCATIONS:
Overall Officials: Youssef BENNIS, MD, Principal Investigator — CHU Amiens; Jean Philippe LANOIX, MD, Study Chair — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No